CLINICAL TRIAL: NCT01886807
Title: The Use of Apneic Oxygenation During Prolonged Intubation in Pediatric Patients: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Peter Szmuk, Professor of Anesthesiology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Apneic Oxygenation
Record Dates: First submitted 2013-06-19; First posted 2013-06-26 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Intubation of Pediatric Dental Surgery Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- (DL group) (Other): direct laryngoscopy for nasotracheal intubation without oxygen insufflation
  Interventions: Device: TrueView PCD Video Laryngoscope
- (DL-O2 Group) (Other): direct laryngoscopy for nasotracheal intubation with oxygen insufflation
  Interventions: Device: TrueView PCD Video Laryngoscope
- (VL Group) (Experimental): nasotracheal intubation using the Truview PCD video laryngoscope
  Interventions: Device: TrueView PCD Video Laryngoscope

INTERVENTIONS:
Device: TrueView PCD Video Laryngoscope

SUMMARY:
Patient demographics (age, height and weight) will be collected for 546 consecutive patients presenting for dental restoration under general anesthesia. The baseline saturation will be recorded. The induction of anesthesia will be standardized for all patients. All patients will undergo an inhalational induction administered by face mask. After inserting an intravenous (IV) line, rocuronium will be administered. Intravenous propofol and fentanyl could be added at the discretion of the anesthesiologist. The patients will be mask ventilated then be with a mixture of Air/Oxygen (O2) to achieve an FiO2 of 0.3 for 3 minutes after the administration of rocuronium.

Patients will be randomly assigned to one of three groups for the purpose of airway management: 1) direct laryngoscopy for nasotracheal intubation without oxygen insufflation (DL group); 2) direct laryngoscopy for nasotracheal intubation with oxygen insufflation (DLO2 Group); and 3) nasotracheal intubation using the Truview PCD video laryngoscope (VL Group). Computer-generated treatment allocations (using the PLAN procedure in SAS statistical software, using random-sized blocks) will be maintained in sequentially numbered sealed envelopes that will be opened after consent is obtained. The laryngoscopy and intubations will be performed by the study investigators who are faculty anesthesiologists or by the mid-level or resident or fellow working with them.

The study will be stopped when:

* the patient will be intubated and a CO2 trace is obtained on the capnography or
* if the patient desaturates to 90%
* or if the patient shows signs of cardiac instability (ectopic beats, arrhythmia or hypotension)

Randomized groups will be compared for balance on potentially confounding baseline variables using descriptive statistics. Primary outcome: In the primary hypothesis, desaturation will be characterized using both time to 1% saturation drop from the baseline and the rate (slope) of desaturation after an initial 1% drop. We will consider a given intubation technique (DLO2 or VL) better than DL on controlling saturation if found noninferior (i.e., not worse) on both outcomes and superior on at least one of the outcomes. Thus our primary hypothesis will be assessed in a joint hypothesis testing framework described by Mascha and Turan. We a-priori define the non-inferiority delta for the outcome time to 1% drop as 5 seconds (or 1.05 if using hazard ratio) and the slope delta as 0.05 percent per second.

DETAILED DESCRIPTION:
Secondary outcomes:

Secondary-1. We will conduct tests for superiority to compare the Truview and DL with oxygen cannula methods on each of the two primary outcomes, and report the treatment effect estimates and adjusted confidence intervals. Notably, the study is not powered to be able to assess equivalence between these two oxygen techniques.

Secondary-2. We will compare the three randomized groups on total desaturation slope (rate) using a random slope linear mixed effects model with repeated measures. This model will allow accounting for the variability of the saturation rate for the patients and possible correlation of the saturation measurements within a patient (autoregressive correlation). We only will use saturation data before it reaches 90%.

Secondary-3. We will assess the relative efficacy of Truview and DL with oxygen cannula in preventing 90% saturation compared with DL alone using 2-tailed chi-square tests of proportions (for superiority), summarized with a relative risk and confidence interval.

Secondary -4: We will assess the correlation between the rate of desaturation and both age and body mass index, independent of randomized group. This will be done in the context of a random slope model as in the primary aim, assessing the interaction between the mean desaturation slope and each of age and body mass index.

To restrict overall Type I error of the secondary hypotheses at 5% we will apply Bonferroni correction for multiple inferences and adjustment for interim analyses.

Interim analyses will be conducted every 25% of the maximum planned enrollment using a groups sequential design to test for efficacy and futility. We will use a gamma spending function (gamma = -4 for efficacy and -2 for futility) to maintain the significance level for the primary outcome at 2.5% and the power at 90% across the interim analyses. Significance criteria for all tests will be adjusted for interim analyses based on the above-mentioned gamma spending function and the corresponding z-statistic at teach interim look.

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for dental restoration under general nasotracheal anesthesia
* Patient age 1-17 years
* American Society of Anesthesiology physical status I, II, III.

Exclusion Criteria:

* Patients at risk of pulmonary aspiration
* Patient with known or suspected difficult airway
* Respiratory infections/disease
* Congenital heart disease
* Hemodynamic instability
* Patients with known latex allergy
* Increased intracranial pressure
* Patients with known or suspected basilar skull fracture
* American Society of Anesthesiology physical status ≥ IV

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 482 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Steiner, DO, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Steiner JW, Sessler DI, Makarova N, Mascha EJ, Olomu PN, Zhong JW, Setiawan CT, Handy AE, Kravitz BN, Szmuk P. Use of deep laryngeal oxygen insufflation during laryngoscopy in children: a randomized clinical trial. Br J Anaesth. 2016 Sep;117(3):350-7. doi: 10.1093/bja/aew186. Epub 2016 Jul 27. PMID 27466252

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | (DL Group) | (DL-O2 Group) | (VL Group)
Started | 164 | 155 | 163
Completed | 159 | 145 | 153
Not Completed | 5 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (DL Group) | (DL-O2 Group) | (VL Group) | Total
Number analyzed (Participants) | 159 | 145 | 153 | 457
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.3 (1.9) | 4.4 (2.1) | 4.7 (2.0) | 4.5 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 71 | 72 | 214
  Male | 88 | 74 | 81 | 243

OUTCOME MEASURES:

1. Primary Outcome: Time of Oxygen Saturation Change
Description: In the primary hypothesis, desaturation will be characterized using both time to 1% saturation drop from the baseline and the rate (slope) of desaturation after an initial 1% drop.We will consider a given intubation technique (DLO2 or VL) better than DL on controlling saturation if found noninferior (i.e., not worse) on both outcomes and superior on at least one of the outcome. From start of intubation attempt to completion of intubation.
Time Frame: From start of intubation attempt to completion of intubation, up to 1 hour
Measure: Mean (95% Confidence Interval); unit: seconds
Groups:
- (DL Group): direct laryngoscopy for nasotracheal intubation without oxygen insufflation
  TrueView PCD Video Laryngoscope
- (DL-O2 Group): direct laryngoscopy for nasotracheal intubation with oxygen insufflation
  TrueView PCD Video Laryngoscope
- (VL Group): nasotracheal intubation using the Truview PCD video laryngoscope
  TrueView PCD Video Laryngoscope
Arm/Group | (DL Group) | (DL-O2 Group) | (VL Group)
Number analyzed (Participants) | 159 | 145 | 153
seconds | 30 [24 to 39] | 67 [35 to 149] | 75 [37 to 122]

2. Primary Outcome: Time to 1% Saturation Drop
Description: Kaplan-Meyer estimate 25th percentile along with adjusted 95% confidence limits were reported instead of usual 50th percentile (median) since there was not enough non-censored data for the DLO2 group (not many patients dropped 1% in SO2 from their baseline )
Time Frame: From beginning to end of laryngoscopy
Measure: Median (95% Confidence Interval); unit: seconds
Arm/Group | (DL Group) | (DL-O2 Group) | (VL Group)
Number analyzed (Participants) | 159 | 145 | 153
seconds | 30 [24 to 39] | 67 [35 to 149] | 75 [37 to 122]

3. Secondary Outcome: Heart Rate
Time Frame: From start of intubation, up to 10 mins
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | (DL Group) | (DL-O2 Group) | (VL Group)
Number analyzed (Participants) | 159 | 145 | 153
beats per minute | 110 (27) | 114 (24) | 110 (26)

4. Secondary Outcome: Systolic Blood Pressure
Time Frame: From start of intubation attempt to completion of intubation, up to 10 mins
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | (DL Group) | (DL-O2 Group) | (VL Group)
Number analyzed (Participants) | 164 | 155 | 163
mmHG | 97 (12) | 98 (14) | 99 (13)

ADVERSE EVENTS:
Arm/Group | (DL Group) | (DL-O2 Group) | (VL Group)
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/155 | 0/163
Other Adverse Events (participants affected / at risk) | 0/164 | 0/155 | 3/163
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (DL Group) (N=164) | (DL-O2 Group) (N=155) | (VL Group) (N=163)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No